CLINICAL TRIAL: NCT05214612
Title: Predictors and Prognostic Factors of Myasthenia Gravis Outcome
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nourelhoda Ahmed Ahmed Haridy, Principal investigator, Lecturer of Neurology, Assiut University
Other Study IDs: Myasthenia gravis Outcome
Record Dates: First submitted 2021-12-31; First posted 2022-01-28 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Myasthenia Gravis; Autoimmune Diseases of the Nervous System; Neuromuscular Junction Diseases; Thymoma; Thymus Hyperplasia; Nervous System Diseases; Myasthenia Gravis, Generalized; Myasthenia Gravis, Ocular; Myasthenia Gravis Crisis; Myasthenia Gravis With Exacerbation (Disorder); Myasthenia Gravis, Adult Form; Myasthenia Gravis, Juvenile Form
Keywords: Predictors; Prognostic factors; Myasthenia Gravis; Outcome
MeSH Terms: conditions — Myasthenia Gravis; Autoimmune Diseases of the Nervous System; Neuromuscular Junction Diseases; Thymoma; Thymus Hyperplasia; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Drug treatment of myasthenia gravis and treatment of crisis — Patients with myasthenia gravis who are receiving medical treatment and treatment of crisis as plasmapheresis

SUMMARY:
This study aims to characterize the clinical features, frequency of different subgroups of MG, and identify predictors of treatment responsiveness among different subgroups of MG. The predictors are including primary outcome (percentage of changes in MG scales at baseline at time of enrollment and after 3 months) and secondary outcome (treatment-related adverse events). Also it aims to determine the frequency of patients with refractory MG.

This information will be used to understand the trends and mechanisms of disease relapse, and optimal management strategies.

DETAILED DESCRIPTION:
Myasthenia gravis (MG) is a rare acquired autoimmune disease affecting the neuromuscular junction (NMJ), caused by autoantibodies that target the post-synaptic membrane. It's overall prevalence ranged from 150 to 250 cases per million. The most common autoantibodies are those directed to the nicotinic acetylcholine receptor (AChR), but there is smaller proportion of cases, in whom, other antibodies can be present and they included antibodies directed to muscle specific tyrosine kinase (MuSK) or to lipoprotein receptor-related protein 4 (Lrp-4). The manifestation of MG is in form of fatigable skeletal muscle weakness, affecting ocular, bulbar and limb muscles. In general, the disease diagnosis is confirmed by presence of this characteristic muscle weakness with positive autoantibodies in the serum. The main current treatment of the disease is symptomatic and immunomodulating therapies which are efficient in managing the disease manifestation. The disease prognosis is mostly favorable and about 15%, is considered medically refractory to the conventional therapy. MG can be classified into different subgroups according to different factors which included the autoantibody status, age of onset, and degree of muscle affection. These subgroups are significantly influencing the therapeutic decisions. Moreover, this proposed classification could explain the distinct immunopathological, clinical, therapeutic, and prognostic differences among these subgroups.

Current standard immunotherapies have a broad-spectrum of immune suppression, and potential side effects associated with their use can significantly impact quality of life, especially as they are usually needed life-long. Significant heterogeneity in treatment responsiveness and outcomes exists among the various subgroups of MG based on epidemiology, clinical presentation, autoantibody status, and comorbidities. In MG clinical trials, the evaluation is mainly depending on the short-term clinical efficacy, but the long-term benefits and impact on patient's quality of life and other disease burdens, (i.e., treatment-related side effects, financial impact), were not measured. The outcomes of MG were assessed in many studies and they included the reduction in quality of life, the negative impact on social and physical health, that related to the disease itself and the immunomodulators used for its treatment. Based on these factors, the investigators aimed to conduct this study to find the disease characteristics in the participants, the patient-tailored targeted treatment strategies, treatment outcomes, disease progression and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 16 years and older.
2. Gender: both sexes are included.
3. Clinical Diagnosis of MG with supporting evidence as:

   1. unequivocal clinical response to pyridostigmine
   2. decrement >10% in repetitive nerve stimulations study (RNS).
4. Willingness to sample collection, imaging study and other disease-related examinations and assessments.

Exclusion Criteria:

1. Age younger than 16 years.
2. History of chronic psychiatric or neurological disorder other than MG that can produce weakness or fatigue.
3. Severe systemic illness affecting life-expectancy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with MG either ocular disease or generalized disease associated with thymoma or not or post-thymectomy, from the outpatient clinics and inpatient wards will be eligible to participate.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in MG-specific Activities of Daily Living scale (MG-ADL). | The changes in points from baseline assessment score to 3 months follow up assessment score
  The MG Activities of Daily Living (MG- ADL) Scale an easily administered, 8-item questionnaire. Each item is graded on a 4- point symptom severity scale (0 = normal, 3 = most severe), with the total score ranging from 0 to 24. Test items emphasize the functional impact of muscle weakness (eg, the ability to comb one's hair or brush one's teeth instead of hand grip or outstretched arm strength tests) rather than its quantitation. The MG-ADL requires no special equipment or training and can be administered in 10 minutes. The MG-ADL test domains include ocular (2 items), oropharyngeal (3 items), respiratory (1 item), and extremity/limb (2 items).
Change in MG quality of life 15 (MG-QOL15). | The changes in points from baseline assessment score to 3 months follow up assessment score
  Everyday clinical use led to the development of an abbreviated 15-item version, the MG-QOL15. These 15 items were derived from the mobility (9 items), symptoms (3 items), general contentment (1 item), and emotional well-being (2 items) domains of the 60-item version. Each of the items/statements (eg, "I have limited my social activity because of my condition") is scored by patients on a 5-point scale ranging from 0 ("not at all") to 4("very much") based on their experience over the previous 4 weeks; the item scores are summed to generate a total score ranging from 0 to 60.
Change in MG manual muscle testing (MG-MMT). | The changes in points from baseline assessment score to 3 months follow up assessment score
  The MG-MMT assesses the strength or function of 30 muscle groups typically affected by MG and includes a total of 18 items, with 12 assessed bilaterally, and 6 assessed as single items (lid closure, cheek puff, tongue protrusion, jaw closure, neck flexion, and neck extension). Each item is scored on a 5- point severity scale, based on the severity of muscle weakness [0 = no weakness, 1 = weak/mild (25%) impairment, 2 = weak/moderate (50%) impairment, 3 = weak/severe (75%) impairment, 4 = paralyzed/unable to perform]. Bilateral scores are summed for a total item score, and all item scores are summed for a total MG-MMT score. MG-MMT scores range from 0 to 120; domains include ocular (3 items, including eyelid closure), facial/oropharyngeal (3 items), axial strength (neck flexion/extension; 2 items), and limb strength (10 items).
Change in MG composite (MGC) Score. | The changes in points from baseline assessment score to 3 months follow up assessment score
  The MG Composite (MGC) Scale is considered a mixed outcome measure that incorporates both physician-evaluated and patient-reported outcome items. In creating this composite scale, the developers sought to minimize the number of items (and thus administration time), to maximize the sensitivity and clinical relevance of each item, and to weight items (as recommended by the Myasthenia Gravis Foundation of America MGFA task force) commensurate with their impact on functional status, QOL, overall health status, and prognosis.13 The MGC Scale is composed of individual items from outcome measures (including the quantitative myasthenia gravis score (QMG), the MG-ADL, and the MG-MMT). Total score spans from 0 to 50.

SECONDARY OUTCOMES:
The proportion of patients with treatment related adverse effects. | At baseline and after 3 months
  Adverse effects of treatment of myasthenia gravis
The proportion of patients reaching minimal manifestations (MM) or better | After 3 months
  Clinical statuses of patients are assessed and categorized according to Myasthenia Gravis Foundation of America (MGFA) postintervention status (PIS). It assesses the clinical state of MG patients at any time after institution of treatment for MG

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gilhus NE. Myasthenia Gravis. N Engl J Med. 2016 Dec 29;375(26):2570-2581. doi: 10.1056/NEJMra1602678. No abstract available. PMID 28029925
- [Background] Sanders DB, Wolfe GI, Benatar M, Evoli A, Gilhus NE, Illa I, Kuntz N, Massey JM, Melms A, Murai H, Nicolle M, Palace J, Richman DP, Verschuuren J, Narayanaswami P. International consensus guidance for management of myasthenia gravis: Executive summary. Neurology. 2016 Jul 26;87(4):419-25. doi: 10.1212/WNL.0000000000002790. Epub 2016 Jun 29. PMID 27358333
- [Background] Evoli A. Myasthenia gravis: new developments in research and treatment. Curr Opin Neurol. 2017 Oct;30(5):464-470. doi: 10.1097/WCO.0000000000000473. PMID 28654435
- [Background] Gilhus NE, Tzartos S, Evoli A, Palace J, Burns TM, Verschuuren JJGM. Myasthenia gravis. Nat Rev Dis Primers. 2019 May 2;5(1):30. doi: 10.1038/s41572-019-0079-y. PMID 31048702
- [Background] Lascano AM, Lalive PH. Update in immunosuppressive therapy of myasthenia gravis. Autoimmun Rev. 2021 Jan;20(1):102712. doi: 10.1016/j.autrev.2020.102712. Epub 2020 Nov 13. PMID 33197578
- [Background] Suh J, Goldstein JM, Nowak RJ. Clinical characteristics of refractory myasthenia gravis patients. Yale J Biol Med. 2013 Jun 13;86(2):255-60. Print 2013 Jun. PMID 23766745
- [Background] Silvestri NJ, Wolfe GI. Treatment-refractory myasthenia gravis. J Clin Neuromuscul Dis. 2014 Jun;15(4):167-78. doi: 10.1097/CND.0000000000000034. PMID 24872217
- [Background] Anil R, Kumar A, Alaparthi S, Sharma A, Nye JL, Roy B, O'Connor KC, Nowak RJ. Exploring outcomes and characteristics of myasthenia gravis: Rationale, aims and design of registry - The EXPLORE-MG registry. J Neurol Sci. 2020 Jul 15;414:116830. doi: 10.1016/j.jns.2020.116830. Epub 2020 Apr 16. PMID 32388060
- [Background] Jaretzki A 3rd, Barohn RJ, Ernstoff RM, Kaminski HJ, Keesey JC, Penn AS, Sanders DB. Myasthenia gravis: recommendations for clinical research standards. Task Force of the Medical Scientific Advisory Board of the Myasthenia Gravis Foundation of America. Ann Thorac Surg. 2000 Jul;70(1):327-34. doi: 10.1016/s0003-4975(00)01595-2. No abstract available. PMID 10921745